CLINICAL TRIAL: NCT03744572
Title: Prestige Pilot - Phoenix Atherectomy and Stellarex DCB Clinical Investigation in Infrapopliteal Interventions
Status: Completed | Type: Observational
Sponsor: Michael Lichtenberg, MD (Other)
Responsible Party: Sponsor-Investigator, Michael Lichtenberg, MD, Chief medical officer Vascular Center, Klinikum Arnsberg
Organization: Klinikum Arnsberg (Other)
Other Study IDs: ASL201801
Record Dates: First submitted 2018-11-04; First posted 2018-11-16 (Actual); Last update posted 2023-01-26 (Actual); Status verified 2023-01

CONDITIONS: Peripheral Artery Disease (PAD)
Keywords: atherectomy; Drug coated balloon
MeSH Terms: conditions — Peripheral Arterial Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This pilot study is to investigate if a lesion preparation strategy with Phoenix atherectomy before DCB (drug coated balloon) usage in patients with PAD (peripheral artery disease) Rutherford Stage 4-5 and mild/moderate/severe calcium can improve outcomes including patency and limb salvage and evaluate safety and performance of the combination therapy

ELIGIBILITY:
Inclusion Criteria:

1. Patients must be ≥ 18 years of age.
2. Patients are male or, if female, are either not of childbearing potential or must have a negative pregnancy test done within 7 days prior-index procedure and effective contraception must be used during participation in the Clinical Investigation.
3. Patients who are mentally and linguistically able to understand the aim of the Clinical Investigation and to show sufficient compliance in following the Clinical Investigation Plan.
4. Patients must agree to return for all required post-index procedure follow-up visits.
5. Patients are able to verbally acknowledge an understanding of the associated risks, benefits, and treatment alternatives to therapeutic options of the Clinical Investigation. Patients, by providing their informed consent, agree to these risks and benefits as stated in the patient informed consent document.
6. Rutherford Class 4-5
7. ≥ 70% stenosis infrapopliteal lesion by angio visual assessment (later correlated with IVUS)
8. Target vessel(s) reconstitute(s) at or above the ankle with inline flow to at least one patent pedal vessel (includes perforating peroneal branches to dorsalis pedis and plantar artery).
9. The target lesion must either be de-novo or restenotic (stenosis ≥ 70% or occlusion by visual estimate). If the target lesion is restenotic, the prior PTA must have been done > 30 days prior-index procedure.
10. Treatment of multiple target lesions is allowed, as long as the composite target lesion length is ≤ 27 cm and the target lesions can be treated with a maximum of 2 overlapping Investigational Devices.
11. Presence of clearly visible calcification in two views (both sides of vessel at the same location) evaluated angiographically- [OPTIONAL: Computerized tomography (CT) angio images may substitute to confirm distribution of calcium, if available as standard of care]
12. Length of calcium ≥ 25 % of total lesion length or ≥ 2 cm total length by angio visual assessment (later correlated with IVUS)
13. At least one target lesion that is ≥ 2cm in length

Exclusion Criteria:

1. Patients with a known hypersensitivity or contraindication to aspirin, heparin, clopidogrel, or other anticoagulant/anti-platelet therapies, Paclitaxel (or analogs) or sensitivity to contrast media that cannot be adequately premedicated.
2. Patients with any contraindications as mentioned in the Instructions for Use (IFU) of the Investigational Device.
3. Patients with a life expectancy, from the Investigator's opinion, of less than 2 years.
4. Patients that are currently participating in other clinical investigations involving any investigational drug or device that may potentially confound the results of the Clinical Investigation, or that would limit the patient's compliance with the follow-up requirements of the Clinical Investigation.
5. Patients with a history of Myocardial Infarction (MI), thrombolysis or angina within 30 days prior-index procedure.
6. Patients with a history of major disabling stroke within 3 months prior index procedure.
7. Patients with any type of previous or planned surgical or interventional procedure within 15 days prior- and/or within 30 days post-index procedure.
8. Patients with a presence or history of severe renal failure (Glomerular Filtration Rate (GFR) ≤ 30 ml/min).
9. Patients who have undergone prior vascular surgery of the index limb to treat atherosclerotic disease.
10. Patients with clinically significant aneurysmal disease of the iliac, femoral or popliteal artery and patients with a history of clinically significant abdominal aortic aneurysm.
11. Treatment of the contralateral limb during the same index procedure or within 30 days post-index procedure in order to avoid confounding complications.
12. Target vessel(s) reconstitute(s) below the ankle with no inline flow to at least one patent pedal vessel.
13. Subjects scheduled to undergo a planned major amputation
14. Prior stent placement in the target lesion(s)
15. Unsuccessful guidewire crossing
16. Subintimal guidewire placement (confirmed by IVUS, no subintimal placement is allowed)
17. Persistent inflow disease left untreated or unsuccessfully treated
18. Non ischemic ulcers and/or ulcers at or above the ankle

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients from clinics with vascular centers
Sampling Method: Probability Sample
Enrollment: 56 (Actual)
Dates: Start 2018-10-17 (Actual); Primary Completion 2020-12-22 (Actual); Study Completion 2022-06-01 (Actual)

PRIMARY OUTCOMES:
Number of target lesions with patency at 6 months | 6 months
  Patency defined as freedom from occluded target lesions (flow) verified by duplex ultrasound without re-intervention
Composite Safety; Number of patients with freedom from BTK major adverse limb events (MALE) and/or perioperative death (POD) | 30-days
  Freedom from BTK major adverse limb events (MALE) and/or perioperative death (POD)

SECONDARY OUTCOMES:
Number of patients with limb salvage | 6, 12, and 24 months
  Limb salvage is defined as freedom from major amputation
Number of target lesions with patency as indicated by PSVR measurement | 6,12, and 24 months
  Patency defined as freedom from >50% restenosis in the target lesion as indicated by a duplex ultrasound peak systolic velocity ratio (PSVR) < 2.5 or by visual assessment of an angiogram with no clinically driven reintervention
Number of target lesions with secondary patency | 6, 12 and 24 months
  Secondary patency is defined as freedom from occluded target lesions (flow) verified by duplex ultrasound
Number of target lesions with procedural success | at end of percutaneous revascularization index procedure
  Procedural sucess is defined as achievement of a ≤30% Diameter Stenosis (DS) at the end of the procedure without MAEs as determined by angiographic core lab
Number of target lesions with technical success | at end of percutaneous revascularization index procedure
  Technical sucess is defined as achievement of a ≤30% Diameter Stenosis (DS) following Phoenix and DCB as determined by angiographic core lab
Number of target lesions with device success for Phoenix atherectomy | during percutaneous revascularization index procedure post-Phoenix and before DCB treatment
  Device success is defined as achievement of a ≤50% Diameter Stenosis (DS) post-Phoenix without pre-dilatation and before DCB or any adjunctive therapy as determined by angiographic core lab
Wound, Ischemia, foot Infection (WIfI) Classification on target limb | 1, 6,12 and 24 months
Ankle-Brachial Index (ABI) | 1, 6,12 and 24 months
Clinical success at follow-up, | 1, 6, 12 or 24 months
  improvement of at least one Rutherford class compared to the pre-procedure Rutherford classification
Pain rating scale scores compared to Baseline | 1, 6, 12 or 24 months
  Pain in the legs during the last 24 h rated on a numerical scale from 0 (no pain) to 10 (worst possible pain)
Walking Impairment Questionnaire (WIQ) score compared to Baseline | 1, 6, 12 or 24 months
  The total WIQ score is defined as sum of five subscores. A subscore is calculated as sum of a scale for each of five separate domains.
Percentage of complete wound healing (complete epithelialization) | 1, 6, 12 or 24 months
correlation between IVUS metrics and angiographic core lab assessment | pre- and at end of percutaneous revascularization index procedure
  Core lab assessed correlation between IVUS metrics of true luminal diameter, actual % area stenosis, change in plaque area and luminal gain pre- and post-therapy, plaque shape and angiographic core lab assessment of pre- and post-percent diameter stenosis (%DS) and the extent of vascular calcification will be determined
Number of patients without Major Adverse Event (MAE) | 6, 12, or 24 months
  MAEs defined as clinically-driven target lesion revascularization, major amputation of the treated limb, and all-cause death

CONTACTS AND LOCATIONS:
Overall Officials: Michael Lichtenberg, Dr., Principal Investigator — Vascular Center, Klinikum Hochsauerland GmbH
Locations (5):
- Germany (5):
  - Vascular Center of Klinikum Hochsauerland, Arnsberg
  - Universitäts-Herzzentrum Bad Krozingen, Bad Krozingen
  - SRH Klinikum Karlsbad-Langensteinbach, Karlsbad
  - St Franziskus Hospital Münster, Münster
  - GRN Klinik Weinheim, Weinheim